CLINICAL TRIAL: NCT06856811
Title: Condylar Position Changes in Anterior Disc Displacement with Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sana'a University (Other)
Responsible Party: Principal Investigator, Suha Hussein Mohammed Almoqayad, condylar position changes in anterior disc displacement with reduction, Sana'a University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: tmj lavage
Record Dates: First submitted 2025-02-24; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: TMJ Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- unilateral anterior disc displacement with reduction (Experimental)
  Interventions: Procedure: tmj lavage with ringer lactate solution

INTERVENTIONS:
Procedure: tmj lavage with ringer lactate solution — tmj lavage using 150ml ringer lactate in symptomatic side of unilateral anterior disc displacement with reduction

SUMMARY:
the goal of this clinical trial is to know if TMJ lavage does change the condyle position in patients diagnosed with unilateral anterior disc displacement with reduction. The main questions it aims to answer are:

* Is the condyle position in anterior disc displacement with reduction joints are the same in normal joints?
* Does TMJ lavage will affect the condyle position, or affects the contralateral condyle position? Researchers will compare condyle position in unilateral anterior disc displacement with reduction to the normal joint using CBCT before and after lavage to see if any changes in position will occur in even side.

Participants will:

Make CBCT for both condyles before lavage and after three months post lavage. Visit clinic after two weeks, one month, and three months to evaluate the clinical data.

ELIGIBILITY:
Inclusion Criteria:

* • Unilateral anterior disc displacement with reduction according to Helkimo's clinical dysfunction index including (Covert et al., 2021a).:

  1. Impaired range of movement.
  2. Impaired TMJ dysfunction.
  3. Muscles pain.
  4. TMJ pain.

Exclusion Criteria:

* • Bilateral anterior disc displacement with reduction.

  * Previous fracture in TMJ.
  * Any pathological lesion in TMJ.
  * Congenital craniofacial anomalies.
  * Any previous surgical procedure in TMJ.
  * Any medically compromised patient (mental deficiency, osteoporosis…)
  * Previous arthrocentesis in TMJ.
  * Partial or complete edentulous patients.
  * Any psychological patient.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
measuring joint spaces in coronal, sagittal and axial views in mm as follows: sagittal view: measuring superior, posterior and anterior space, coronal measuring medial and lateral joint spaces, axial measuring the intercondylar distance and angle | three months follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Sana'a University, Sanaa, Yemen